CLINICAL TRIAL: NCT06612164
Title: Effects of Kefir Consumption on Health Outcomes: Gastrointestinal System, Immunity, Biochemical Parameters, Body Composition, Sleep Quality and Mental Well Being in Healthy Adults
Acronym: KefirCons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Merve Pehlivan, PhD, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 720
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Effect of Kefir on Healthy Adults
Keywords: gastrointestinal symptoms; immunity; kefir; mental health; sleep quality; body composition
MeSH Terms: conditions — Psychological Well-Being; Sleep Initiation and Maintenance Disorders | interventions — Kefir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kefir Consumption Group (Experimental): Commercial lactose-free kefir (Altinkilic, Turkey) beverage, which is produced from cow milk with 3.1% fat and 7.5% protein content and stored in appropriate conditions, was used in this study. The kefir (intervention) group was provided with 250 mL of plain lactose-free kefir containing at least 107-1010 probiotic bacterial strains (Lactobacillus, Lactic acid, Streptococcus, Acetic acid bacteria sp) and yeasts (Kluyveromyces marxianus, Torulaspora delbrueckii, Saccharomyces cerevisiae, Candida). The participants were asked to consume 250 mL of plain lactose-free kefir daily for 6 weeks. Any particular time was not specified for kefir consumption. Kefir consumption routine of participants was followed up by regular phone calls every week and evaluated by examining their consumption records.
  Interventions: Other: kefir
- Control Group (No Intervention): Short Physical Activity Assessment Tool was used for evaluating physical activity levels of the participants, mental health status by The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Gastrointestinal system symptoms were evaluated by using the Gastrointestinal Symptom Rating Scale (GSRS), sleep quality by the Pittsburg Sleep Quality Index (PSQI) and diet quality by the Healthy Eating Index-2015 (HEI-2015). Measurements were recorded prior to kefir intervention (initial measurement) and post kefir intervention (final measurement) for kefir and control groups.

INTERVENTIONS:
Other: kefir — Commercial lactose-free kefir (Altinkilic, Turkey) beverage, which is produced from cow milk with 3.1% fat and 7.5% protein content and stored in appropriate conditions, was used in this study. The kefir (intervention) group was provided with 250 mL of plain lactose-free kefir containing at least 107-1010 probiotic bacterial strains (Lactobacillus, Lactic acid, Streptococcus, Acetic acid bacteria sp) and yeasts (Kluyveromyces marxianus, Torulaspora delbrueckii, Saccharomyces cerevisiae, Candida). The participants were asked to consume 250 mL of plain lactose-free kefir daily for 6 weeks. Any particular time was not specified for kefir consumption. Kefir consumption routine of participants was followed up by regular phone calls every week and evaluated by examining their consumption records. Those who consumed less than 85.0% (skipping kefir consumption maximum once a week) of the planned kefir consumption during the study period were excluded from the study.
  Arms: Kefir Consumption Group

SUMMARY:
The goal of this clinical trial is to evaluate the effects of the administration of kefir on gastrointestinal system, mental health, biochemical parameters, immunity and inflammation processes as well as the sleep quality, elucidating the possible health effects of kefir consumption in healthy adults. The main questions it aims to answer are:

1. Will be better the gastrointestinal system symptoms severity of volunteers in the intervention group will be better compared to the control group?
2. Will be better the mental health status of volunteers in the intervention group will be better compared to the control group?
3. Will be better the biochemical parameters of volunteers in the intervention group will be better compared to the control group?
4. Will be better the immunity and inflammation processes of volunteers in the intervention group will be better compared to the control group?

The participants were asked to consume 250 mL of plain lactose-free kefir daily for 6 weeks. Any particular time was not specified for kefir consumption. Kefir consumption routine of participants was followed up by regular phone calls every week and evaluated by examining their consumption records. Those who consumed less than 85.0% (skipping kefir consumption maximum once a week) of the planned kefir consumption during the study period were excluded from the study.

DETAILED DESCRIPTION:
In order to evaluate the general characteristics, history of diseases and nutritional behaviors, a face-to-face questionnaire was conducted on all participants by the researchers. The questionnaire form contained information about the demographic information (age, gender, educational status, marital status, etc.), history of diseases (diagnosed diseases, drugs used etc.), basic nutritional habits (number of major meals/snacks consumed in a day, water consumption, etc.) and anthropometric measurements (body weight, height, body mass index, waist circumference, neck circumference). In the intial (pre-intervention) and final (post-intervention) stages of the study, anthropometric measurements of the participants were taken, and body composition analysis was done. In addition, biochemical findings and 3-day food consumption records were taken in the intial (pre-intervention) and final (post-intervention) stages of the study. Effects of kefir consumption on gastrointestinal system, biochemical findings, mental health, immunity and inflammation, sleep quality, was evaluated by assessment of the relevant status of participants before and after kefir intervention and comparison with the control group. Short Physical Activity Assessment Tool was used for evaluating physical activity levels of the participants, mental health status by The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Gastrointestinal system symptoms were evaluated by using the Gastrointestinal Symptom Rating Scale (GSRS), sleep quality by the Pittsburg Sleep Quality Index (PSQI) and diet quality by the Healthy Eating Index-2015 (HEI-2015). Measurements were recorded prior to kefir intervention (initial measurement) and post kefir intervention (final measurement) for kefir and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to consume 250 mL of plain lactose-free kefir once a day,
* Being healthy
* Being 18-35 years of age.

Exclusion Criteria:

* Follow a special diet for health reasons,
* Have an allergy to any food, have hepatic, renal and biliary diseases, have immunodeficiency, autoimmune and chronic gastrointestinal diseases, have a history of cancer, diabetes or cardiovascular diseases,
* Being pregnant/breastfeeding,
* Using vitamin-mineral and probiotic supplements,
* Using antibiotics in last one month and throughout the study period,
* Consuming probiotic foods or kefir on a regular basis,
* Smoking

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Gastrointestinal Health | From enrollment to the end of treatment at 6 weeks
  Gastrointestinal Symptom Rating Scale developed by Revicki et al and validated in Turkish by Turan et al. (2017) was used to evaluate gastrointestinal health of participants. GSRS is a disease specific instrument comprising of 15 items combined into 5 symptom clusters namely abdominal pain (items 1, 4 and 5), reflux (items 2 and 3), indigestion (items 6, 7, 8 and 9), diarrhea (items 11,12 and 14) and constipation (items 10, 13 and 15). In order to score the items, participants state how he/she felt about these problems in the past week. GSRS questions are rated on a 7-point Likert scale ranging from "no discomfort" to "very severe discomfort". A score of 1 is given for the absence of symptoms, and 7 for frequent and severe symptoms. High scores indicate severity of symptoms and diseased state.
Body Composition and Anthropometric Measurements | From enrollment to the end of treatment at 6 weeks
  Body composition analysis, of the participants, was performed with TANITA MC-780 body composition analyser. By means of bioelectrical impedance analysis, basal metabolic rate and body composition (fat mass, muscle mass, fluid mass, lean mass, bone mineral mass, visceral fat, phase angle and edema index) were evaluated. Height (with SECA 206), body weight (with TANITA MC-780), neck and waist circumferences (with SECA 201) of participants were recorded. Heights were measured while standing upright and without shoes, feet were placed side by side, head was placed on the Frankfort Horizontal Plane, occipital region toucing the stadiometer. The body mass index (BMI) of the participants was calculated by dividing the body weight (kg) by the square the height (metres) and the evaluation was made according to the classification of the World Health Organization.
Mental Health | From enrollment to the end of treatment at 6 weeks
  The Warwick-Edinburgh Mental Well-Being Scale developed by Tennant et al. (2007) and validated in Turkish by Keldal (2015), was used to evaluate the mental health status of individuals. The WEMWBS total score is calculated by adding the scores assigned to each of the 14 items (1=never to 5=always). The minimum score that can be obtained is 14, whereas the maximum score obtained is 70. Higher scores are associated with higher mental well-being.
Immunity and Systemic-Inflammation | From enrollment to the end of treatment at 6 weeks
  Evaluation of immunity and systemic inflammation was performed using complete blood cell count and the SII, which is an important marker in reflecting inflammation and immune response. Although platelet-lymphocyte ratio (PLR) and neutrophil-lymphocyte ratio (NLR) are associated with disease activity, however, it has been suggested that SII, which is calculated by using platelet, neutrophil, and lymphocyte counts together, is a much more important marker in showing inflammation and immune response as compared to PLR and NLR values alone. Furthermore, SII is associated with various diseases such as cancer and cardiovascular disease. SII value is calculated with a formula (SII=P×N/L, P; platelet, N; neutrophil, L; lymphocyte) and high scores are associated with adverse health outcomes.

SECONDARY OUTCOMES:
Physical Activity | From enrollment to the end of treatment at 6 weeks
  Participants were asked to maintain their usual physical activities. The physical activity levels of the participants were evaluated with the Short Physical Activity Assessment Tool. The tool consisted of two questions focusing on 20 minutes of vigorous physical activity (running, weightlifting, cycling, etc.) and 30 minutes of moderate physical activity (mowing grass, lifting light loads, etc.). A maximum score of 8 and a minimum score of 0 could be obtained by this tool. A total score of 0-3 was considered insufficiently active, and a score of ≥4 was considered sufficiently active.
Biochemical Parameters | From enrollment to the end of treatment at 6 weeks
  Blood analysis for the following parameters (fasting blood glucose, high density lipoprotein cholesterol (HDL), low density lipoprotein cholesterol (LDL), total cholesterol, triglyceride, alanine transaminase (ALT), aspartate transaminase (AST), blood urea nitrogen (BUN), urea, uric acid, creatinine, bilirubin, C-reactive protein (CRP), iron, iron binding capacity) was performed and the hemogram obtained at the beginning and end (pre and post intervention) of the study. The systemic immune-inflammation index (SII) was calculated from the hemogram findings.
Dietary Patterns | From enrollment to the end of treatment at 6 weeks
  Participants were asked to maintain their usual eating habits. They were asked to record 24-hour food consumption for three non-consecutive days, one of which was required to be a weekend. This food record was taken twice; once at the beginning (prior to kefir intervention) and the other at the end (post kefir intervention) of the study. The records were collected from the participants retrospectively. The average daily energy and nutrient intakes of the individuals were determined by taking the average of the food consumption consumption values of the three days. The dietary quality of the participants was evaluated with the HEI-2015, which was calculated using data from food consumption records. If the HEI-2015 score of the participants was ≤50 points, the diet quality was evaluated as "poor diet quality", 51-80 points as "diet quality to be improved", and >80 points as "good diet quality".

OTHER OUTCOMES:
Sleep Quality | From enrollment to the end of treatment at 6 weeks
  Pittsburg Sleep Quality Index , developed by Buysse et al. (1989) and validated in Turkish by Ağargün et al. (1996), was used to assess sleep quality.. The tool comprises of 7 sub-components and 18 items, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction. The total score is calculated by evaluating the sub-components of the scale over 0-3 points. A score of 0-4 indicates good sleep quality, and a total score of 5-21 points indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bakirhan H, Ozyurek Arpa F, Pehlivan M, Kalkan I. Effects of Kefir Consumption on Gastrointestinal Health, Biochemical Parameters, Sleep, and Mental Well-Being in Healthy Young Adults: a Randomized Controlled Trial. J Nutr. 2026 Jan;156(1):101247. doi: 10.1016/j.tjnut.2025.11.016. Epub 2025 Nov 26. PMID 41314291